CLINICAL TRIAL: NCT00126087
Title: Potentiation of Procedural Motor Learning by Pharmacological Neuromodulation and Transcranial Direct Current Stimulation in Health and Disease
Brief Title: Potentiation of Procedural Motor Learning in Health and Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no further funding available for recruiting and testing participants
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Motor-Neuromod_01
Record Dates: First submitted 2005-07-31; First posted 2005-08-02 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Stroke
Keywords: dopamine; NMDA receptor; brain imaging; neuroplasticity; learning; transcranial direct current stimulation; rehabilitation; aging
MeSH Terms: conditions — Stroke | interventions — Dopamine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: dopamine

SUMMARY:
The investigators plan to improve the learning of motor skills by pharmacological means (dopamine), and by noninvasive brain stimulation. They will study both healthy subjects and chronic stroke patients. In addition, they want to study the mechanisms of enhanced learning, on the molecular and the systems level.

DETAILED DESCRIPTION:
Adaptive behavior requires procedural motor learning, i.e. the acquisition of motor skills. Procedural learning is particularly critical in the rehabilitation of chronic motor deficits after stroke. A potent modulator of motor function and learning is found in the endogenous dopaminergic system. The investigator's own work could demonstrate that formation of an elementary motor memory, which constitutes the first step in acquiring more complex motor skills, can be enhanced in both healthy subjects and chronic stroke patients by pre-medication with levodopa. The aim of the present proposal is to:

* expand these exciting findings to procedural motor learning;
* explore the interaction with age, brain lesions, add-on interventions such as transcranial direct current stimulation (tDCS); and
* illuminate the underlying mechanisms.

The effect of levodopa +/- tDCS on procedural motor learning and cortical excitability will be studied in healthy volunteers and stroke patients. Then the investigator plans to delineate the underlying mechanisms of this effect by exploring N-methyl-D-asparate (NMDA) receptor-dependency of levodopa-enhanced learning and changes in activation and connectivity (using functional magnetic resonance imaging) in the respective neural networks resulting from the interaction of learning and dopaminergic neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* Normal neurological examination
* Mini Mental State Examination of > 27
* Right handedness

Stroke Patients:

* Cortical or subcortical stroke with an initial severe hemiparesis Medical Research Council (MRC) scale < 2 that has recovered to a degree that patients are able to perform the proposed task (in general > MRC 4.5, with low spasticity, work in progress on motor learning in stroke patients)
* At least 1 year post-stroke
* Mini Mental State Examination of > 27
* Right-handedness

Exclusion Criteria:

Healthy Volunteers and Stroke Patients:

* No antipsychotic, antidepressant drugs, and drugs affecting the dopaminergic system.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Procedural motor learning (decrease in reaction time in ms) after the respective intervention (dopamine, transcranial direct current stimulation), compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, MD, Principal Investigator — University of Münster, Department of Neurology, Germany
Locations (1):
- University of Münster, Department of Neurology, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Floel A, Breitenstein C, Hummel F, Celnik P, Gingert C, Sawaki L, Knecht S, Cohen LG. Dopaminergic influences on formation of a motor memory. Ann Neurol. 2005 Jul;58(1):121-30. doi: 10.1002/ana.20536. PMID 15984008
- [Result] Rosser N, Heuschmann P, Wersching H, Breitenstein C, Knecht S, Floel A. Levodopa improves procedural motor learning in chronic stroke patients. Arch Phys Med Rehabil. 2008 Sep;89(9):1633-41. doi: 10.1016/j.apmr.2008.02.030. PMID 18760148